CLINICAL TRIAL: NCT00458276
Title: Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Efficacy, Safety and Tolerability of Tezosentan in Patients With Pre-operative Pulmonary Hypertension, Due to Left Heart Disease, Undergoing Cardiac Surgery
Brief Title: Study of the Efficacy and Safety of Tezosentan in Patients With Pre-operative Pulmonary Hypertension, Due to Left Heart Disease, Undergoing Open Heart Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: 6 month vital status report not collected after 28 day follow up analysis indicated no difference between placebo & tezosentan
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AC-051-350
Record Dates: First submitted 2007-04-06; First posted 2007-04-10 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Heart Diseases; Hypertension, Pulmonary
Keywords: Left sided heart disease; Elevated pulmonary arterial pressure; Right ventricular failure; Cardiac surgery; heart-lung machine; cardiopulmonary bypass; tezosentan; Actelion
MeSH Terms: conditions — Heart Diseases; Hypertension, Pulmonary; Heart Failure | interventions — tezosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Tezosentan
  Interventions: Drug: tezosentan
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tezosentan — Tezosentan (ACT-050089, Ro 61-0612) as a 1% solution in 0.9% NaCl (i.e., normal saline) for i.v. use.
  Arms: 1
Drug: placebo — Placebo (i.e., normal saline) for i.v. use.
  Arms: 2

SUMMARY:
Endothelin-1 is a powerful substance that may be involved in causing hemodynamic instability (problems related to unstable blood pressure) during and after open heart surgery. Tezosentan is an investigational intravenous drug that blocks the endothelin receptors. This clinical trial will assess the potential benefit of tezosentan compared with placebo in the treatment of patients undergoing open heart surgery with cardiopulmonary bypass (CPB). Treatment time is from the start of surgery up to 24 hours.

DETAILED DESCRIPTION:
Endothelin-1 levels are increased during and after cardiac surgery with cardiopulmonary bypass (CPB), and are associated with many deleterious consequences, including increased pulmonary arterial pressure (PAP), increased pulmonary vascular resistance (PVR), reduced myocardial contractility, and ultimately right ventricular failure. Right ventricular failure during weaning from CPB increases the risk of mortality and morbidity, especially in patients with elevated PAP prior to cardiac surgery. Endothelin receptor antagonists (ERAs) have been shown to decrease PVR and pulmonary arterial pressure (PAP), and improve right ventricular function in patients with pulmonary arterial hypertension. In animal models, ERAs have been shown to decrease the incidence of post-bypass pulmonary hypertensive crises. The primary objective of this trial is to demonstrate that tezosentan, a dual ERA, reduces the incidence of clinically relevant right ventricular failure in patients with pre-operative pulmonary hypertension, due to left heart disease, undergoing CPB.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Male or female patients (females of child-bearing potential must have been surgically sterilized or use a reliable method of contraception).
* Patients undergoing complex* cardiac surgery on CPB and having systolic PAP > 40 mmHg or mean PAP > 30 mmHg (*surgery on 2 valves, 1 valve and revascularization, or reoperation of a valve)
* Patients undergoing cardiac surgery on CPB and having pre-operative pulmonary hypertension due to left heart disease with systolic PAP > 60 mmHg
* Signed written informed consent

Exclusion Criteria:

* Systolic blood pressure < 100 mmHg
* Significant chronic lung disease
* Emergency surgery
* Pregnant/breast-feeding
* Investigational drug use within 28 days prior to randomization
* Complex adult congenital heart disease.
* Severe concomitant illness limiting life expectancy to < 6 months
* Participation in a device study that will affect the outcome of the study
* Pre-operative use of balloon pump, inotropes/vasopressors, treatment of pulmonary arterial hypertension
* Known hypersensitivity to tezosentan or drugs of the same class, or any of their excipients
* Severe liver impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2007-04; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of this trial is to demonstrate that tezosentan, a dual ERA, reduces the incidence of clinically relevant right ventricular failure in patients with pre-operative pulmonary hypertension, due to left heart disease, undergoing CPB. | During weaning from CPB

SECONDARY OUTCOMES:
Proportion of patients w/a major clinical event w/in 28 days after study drug initiation like death/major cardiovascular events/infections that prolong hospital stay or require re-admission/new onset of renal failure requiring renal replacement therapy | Within 28 days after study initiation
Time to weaning from cardiopulmonary bypass | Defined as time from release of cross-clamp to successful weaning from CPB
Time from end of CPB to final discharge from Intensive Care Unit (ICU) | From end of CPB to final discharge from ICU

CONTACTS AND LOCATIONS:
Overall Officials: Andre Denault, Prof., Study Chair — Montreal Heart Institute; Ronald Pearl, MD, Study Chair — Stanford University; Robert Michler, MD, Study Chair — Montefiore Medical Center; Steven Tsui, Study Chair — Papworth Hospital NHS Foundation Trust; Rainald Seitelberger, Prof., Study Chair — AKH University of Vienna; Andrea D'Armini, Prof., Study Chair — San Matteo Hospital
Locations (33):
- United States (9):
  - Stanford University School of Medicine, Stanford, California
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center/Albert Einstein College of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
  - Baylor University Medical Center, Dallas, Texas
  - Texas Heart Institute/St. Luke's Episcopal Hospital/Baylor College, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
- Austria (2):
  - Medical University of Innsbruck, Innsbruck
  - AKH University of Vienna, Vienna
- Canada (5):
  - University of Alberta Hospital, Edmonton, Alberta
  - London Health Sciences Centre-University Hospital, London, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Quebec Heart Institute/Hopital Laval, Québec, Quebec
- Institute for Clinical and Experimental Medicine (IKEM), Prague, Czechia
- Hopital Pitie Salpetriere, Paris, France
- Germany (3):
  - Deutches Herzzentrum, Berlin
  - Dresden Universitatsklinik/Cardiology Center, Dresden
  - Zentrum der Chirugie-Zchir-des Universitatsklinikums, Frankfurt
- India (2):
  - Narayana Hrudayalaya, Bangalore
  - Nizam's Institute of Medical Sciences, Hyderabaad
- Shaare Zedek Medical Center, Jerusalem, Israel
- Italy (2):
  - Fondazione IRCCS San Matteo Hospital, Cardiac Surgery, Pavia
  - Azienda Sanitaria Ospedaliera "San Giovanni Battista", Cardiac Surgery Division, Torino
- Poland (2):
  - Medical University of Silesia, 2nd Dept of Cardiac Surgery, Katowice
  - Klinika Chirurgii Serca, Naczyn I Transplantologii, Szpital Jana Pawla II, Krakow
- Dedinje Cardiovascular Institute, Belgrade, Serbia
- National Institute of Cardiovascular Diseases, Clinic of Heart Surgery, Bratislava, Slovakia
- Sahlgrenska University Hospital, Gothenburg, Sweden
- United Kingdom (2):
  - Papworth Hospital, Cambridge
  - Northern General Hospital, Sheffield

REFERENCES:
- [Derived] Denault AY, Pearl RG, Michler RE, Rao V, Tsui SS, Seitelberger R, Cromie M, Lindberg E, D'Armini AM. Tezosentan and right ventricular failure in patients with pulmonary hypertension undergoing cardiac surgery: the TACTICS trial. J Cardiothorac Vasc Anesth. 2013 Dec;27(6):1212-7. doi: 10.1053/j.jvca.2013.01.023. Epub 2013 Mar 21. PMID 23523254